CLINICAL TRIAL: NCT01673581
Title: Shared Decision Making: A Study Assessing the Benefit of a Web Based Aid Presenting Treatment Options for Patients With Low Risk Prostate Cancer
Brief Title: Shared Decision Making in Low Risk Prostate Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jason Efstathiou, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 11-463
Record Dates: First submitted 2012-08-15; First posted 2012-08-28 (Estimated); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Prostate Cancer
Keywords: Low Risk
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Low risk prostate cancer
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey

SUMMARY:
This study will evaluate the usefulness of an informational website designed to educate patients with prostate cancer about their options for treatment. The investigators hope that this website will assist patients with making informed decisions about their care and improving their satisfaction with the treatments they choose.

DETAILED DESCRIPTION:
Investigators will first ask patients to answer a series of questions to assess their wishes regarding treatment, knowledge about their disease and discussion with the physicians at initial patient visit. This initial survey should take approximately 20 minutes. Once patients have selected a treatment path investigators will contact them again and ask them to fill out a short 10-minute survey online or by mail. Investigators will contact patients by phone 2 weeks after their initial visit to see if they have made a decision. If not, investigators will contact patients by phone every 2 weeks or at an interval that works for the patient's schedule. Finally, 3 months after the initial visit today investigators will contact patients for the last time and again ask you to fill out a short 10-minute survey online or by mail.

Once patients have completed the final survey there are no future surveys planned. Investigators may contact patients by phone in the future to ask them to participate in another study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate adenocarcinoma
* Internet access
* Able to read and understand English

Exclusion Criteria:

* Evidence of nodal metastases
* Evidence of distant metastases
* Prior surgery, chemotherapy, pelvic radiation or prostate brachytherapy for prostate cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Low risk prostate cancer patients seen wthin the Claire & John Bertucci Center for Genitourinary Cancers multidisciplinary clinic at MGH.
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2012-08; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Patient knowledge regarding the available treatment options for low-risk prostate cancer and their potential side effects. | 2 years
  Investigators will assess the impact of an informational website developed specifically to assist low-risk prostate cancer patients with knowledge of their disease and treatment options. This will be measured by patient responses to questionnaires compiled from validated sources.

SECONDARY OUTCOMES:
Decisional conflict and informed decision making experienced by patients. | 2 years
  Investigators will assess the impact of an informational website developed specifically to assist low-risk prostate cancer patients with knowledge of their disease and treatment options. This will be measured by patient responses to questionnaires compiled from validated sources.
Patient health related worry. | 2 years
  Investigators will assess the impact of an informational website developed specifically to assist low-risk prostate cancer patients with knowledge of their disease and treatment options. This will be measured by patient responses to questionnaires compiled from validated sources.
Patient views on cancer control for their treatment choice. | 2 years
  Investigators will assess the impact of an informational website developed specifically to assist low-risk prostate cancer patients with knowledge of their disease and treatment options. This will be measured by patient responses to questionnaires compiled from validated sources.
Patient satisfaction with their treatment choice. | 2 years
  Investigators will assess the impact of an informational website developed specifically to assist low-risk prostate cancer patients with knowledge of their disease and treatment options. This will be measured by patient responses to questionnaires compiled from validated sources.

CONTACTS AND LOCATIONS:
Overall Officials: Jason A. Efstathiou, MD, DPhil, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States